CLINICAL TRIAL: NCT06024798
Title: Assessing Patients With Suspected Stress or Insufficiency Fracture of the Lower Extremity With Photon-Counting-Computed-Tomography
Brief Title: Detecting and Assessing Leg and Foot Stress Fractures Using Photon Counting CT
Acronym: FootPCCT
Status: Recruiting | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: W1024
Record Dates: First submitted 2023-08-21; First posted 2023-09-06 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Stress Fracture Foot; Stress Fracture Ankle; Stress Fracture of Tibia; Stress Fracture Metatarsal; Lower Limb Fracture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 13 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Photon-Counting-Computed-Tomography — Initial and follow up (after 4 weeks) PCCT acquisition of the affected area of the lower extremity. Image acquisition will be performed on the PCCT

SUMMARY:
Stress fractures (fatigue or insufficiency fracture) are caused by the mismatch between bone strength and chronic stress applied to the bone. The vast majority of these fractures occur in the lower extremity. Early-stage diagnosis is crucial to optimize patient care. Appropriate imaging is relevant in confirming diagnosis after clinical suspicion of stress fractures. Radiographs have low sensitivity, so a relevant number of fractures go undetected. MRI has a high sensitivity, but its availability is limited, and its respective examination time is prolonged. This study investigates the diagnostic accuracy of PCCT in lower extremity stress fractures as a dose-saving technology, guaranteeing an examination according to the ALARA-principle (as low as reasonably achievable).

DETAILED DESCRIPTION:
Stress fracture is caused by the mismatch between bone strength and chronical stress applied to the bone, which is insufficient to cause an acute fracture, but a stress fracture does not heal itself. One can subclassify it into fatigue fracture (overuse of a healthy bone) and insufficiency fracture (normal use of a weakened bone). Fatigue fractures usually happen in healthy athletes or military recruits, whereas insufficiency fracture appear in patients with underlying metabolic or nutritional disorder (e.g. osteoporosis). On radiographs and Computed Tomography (CT), stress fractures are defined as round or linear intracortical lucency or an intertrabecular sclerotic line, which rarely intersects the cortex. Radiograph is a cost-effective and highly available modality in detecting fractures, showing however a moderate sensitivity in detecting stress fractures: 15-35% on the initial and 30-70% on the follow-up imaging. CT, another modality highly available in most hospital settings, shows a similar moderate sensitivity of 32-38% with however a corresponding high specificity of 88-98% on initial imaging. Similar specificity values can be observed for magnetic resonance imaging (MRI) and nuclear scintigraphy. Although their availability is limited and their respective examination time is prolonged, they outperform the x-ray based technologies in term of sensitivity (68-98% MRI and 50-97% nuclear scintigraphy, respectively).

The introduction of dual-energy technology advanced CT from a pure anatomical evaluation tool to a combined anatomical and functional modality. Every material has a specific absorption number, which can be assessed by applying two different energies (high and low x-ray tube voltages). This method of multispectral imaging has been established and clinically implemented in detecting gout and characterizing renal stones. Further studies have shown that DECT can depict bone marrow edema, a marker of early stress fracture and a common finding in MRI. However, this has yet not been implemented in clinical practice.

The photon-counting-computed-tomography (PCCT) has been introduced recently, enabling an energy dependent separation of photons over the whole x-ray energy spectrum. This results in reduced background noise, improved image resolution and multispectral imaging without the necessity of an additional acquisition at a different energy level. An initial study has shown already shown the superiority of PCCT by better detecting and characterizing small renal stones, when compared to conventional dual-energy computed tomography (DECT).

In this project the investigators aim to include clinically referred patients with suspected stress fracture of the lower extremity who will have an MRI to confirm the diagnosis of a suspected stress fracture. The subjects will be scanned on the new PCCT system with dose saving technology, guaranteeing an examination according to the ALARA-principle (as low as reasonably achievable). The investigators will not inject iodine contrast media and they will expect a median dose of 2-4 mSv (millisieverts). Since this will not exceed the threshold of 5 mSv, this project will be classified as category A.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 16 years of age. Minor study subjects can have an additional signature by the parent or legal guardian
* Clinically suspected stress or insufficiency fracture of the lower extremity
* Written consent of study participation
* Patients who will have an MRI to confirm the diagnosis of a suspected stress fracture

Exclusion Criteria:

* < 16 years of age
* Pregnancy
* Metal implants
* Postoperative situation
* Infection or tumorous disease affecting the lower extremity

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In cooperation with the Foot Clinic at the Balgrist University Hospital Zurich, potential study candidates with suspected stress fracture who will undergo an MRI to confirm the diagnosis are prospectively screened and proposed to join the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Presence of a fracture | Day 1, 4weeks follow up assessment
  Presence/absence of a fracture

SECONDARY OUTCOMES:
Presence of bone edema | Day 1, 4weeks follow up assessment
  Presence/absence of bone edema
Presence of soft tissue edema | Day1, 4weeks follow up assessment
  Presence/absence of soft tissue edema

OTHER OUTCOMES:
Pain localization | Day 1, 4 weeks follow up assessment, 12 weeks follow up assessment
  Pain localization will be done through a clear statement of anatomical location
Pain character | Day 1, 4 weeks follow up assessment, 12 weeks follow up assessment
  Pain will be characterized using the following terms: sharp, dull, aching, burning, radiating, numbing, and pulsating.
Pain intensity | Day 1, 4 weeks follow up assessment, 12 weeks follow up assessment
  Pain intensity will be described using the Number Rating Scale (NRS): a score of 0 corresponds to the absence of pain, while a score of 10 indicates the most intense pain ever experienced.
Pain duration | Day 1, 4 weeks follow up assessment, 12 weeks follow up assessment
  Pain duration is described in days (d).
Karlsson Scoring Scale: Patient reported outcome regarding the stress fracture | Day 1, 4 weeks follow up assessment, 12 weeks follow up assessment
  The Karlsson scoring scale is utilized to evaluate and quantify both the functional status and the extent to which the stress fracture affects an individual's quality of life. The scoring system comprises a total of 90 points, where 0 points represent the most severe condition and 90 points indicate an absence of any issues.
Foot Function Index: Patient reported outcome regarding the stress fracture | Day 1, 4 weeks follow up assessment, 12 weeks follow up assessment
  The Foot Function Index is utilized to evaluate and quantify both the functional status and the extent to which the stress fracture affects an individual's quality of life. The minimum score is 0% (no pain or difficulty), and maximum score is 100%

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Wirth, PD Dr.med., Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palmer W, Bancroft L, Bonar F, Choi JA, Cotten A, Griffith JF, Robinson P, Pfirrmann CWA. Glossary of terms for musculoskeletal radiology. Skeletal Radiol. 2020 Jul;49(Suppl 1):1-33. doi: 10.1007/s00256-020-03465-1. Epub 2020 Jun 2. PMID 32488336
- [Background] Lassus J, Tulikoura I, Konttinen YT, Salo J, Santavirta S. Bone stress injuries of the lower extremity: a review. Acta Orthop Scand. 2002 Jun;73(3):359-68. doi: 10.1080/000164702320155392. PMID 12143987
- [Background] Wright AA, Hegedus EJ, Lenchik L, Kuhn KJ, Santiago L, Smoliga JM. Diagnostic Accuracy of Various Imaging Modalities for Suspected Lower Extremity Stress Fractures: A Systematic Review With Evidence-Based Recommendations for Clinical Practice. Am J Sports Med. 2016 Jan;44(1):255-63. doi: 10.1177/0363546515574066. Epub 2015 Mar 24. PMID 25805712
- [Background] Wortman JR, Uyeda JW, Fulwadhva UP, Sodickson AD. Dual-Energy CT for Abdominal and Pelvic Trauma. Radiographics. 2018 Mar-Apr;38(2):586-602. doi: 10.1148/rg.2018170058. PMID 29528816
- [Background] Cabarrus MC, Ambekar A, Lu Y, Link TM. MRI and CT of insufficiency fractures of the pelvis and the proximal femur. AJR Am J Roentgenol. 2008 Oct;191(4):995-1001. doi: 10.2214/AJR.07.3714. PMID 18806133
- [Background] Gosangi B, Mandell JC, Weaver MJ, Uyeda JW, Smith SE, Sodickson AD, Khurana B. Bone Marrow Edema at Dual-Energy CT: A Game Changer in the Emergency Department. Radiographics. 2020 May-Jun;40(3):859-874. doi: 10.1148/rg.2020190173. PMID 32364883
- [Background] Grunz JP, Sailer L, Lang P, Schule S, Kunz AS, Beer M, Hackenbroch C. Dual-energy CT in sacral fragility fractures: defining a cut-off Hounsfield unit value for the presence of traumatic bone marrow edema in patients with osteoporosis. BMC Musculoskelet Disord. 2022 Jul 29;23(1):724. doi: 10.1186/s12891-022-05690-2. PMID 35906573
- [Background] Henes FO, Nuchtern JV, Groth M, Habermann CR, Regier M, Rueger JM, Adam G, Grossterlinden LG. Comparison of diagnostic accuracy of Magnetic Resonance Imaging and Multidetector Computed Tomography in the detection of pelvic fractures. Eur J Radiol. 2012 Sep;81(9):2337-42. doi: 10.1016/j.ejrad.2011.07.012. Epub 2011 Sep 15. PMID 21924851
- [Background] Bongartz T, Glazebrook KN, Kavros SJ, Murthy NS, Merry SP, Franz WB 3rd, Michet CJ, Veetil BM, Davis JM 3rd, Mason TG 2nd, Warrington KJ, Ytterberg SR, Matteson EL, Crowson CS, Leng S, McCollough CH. Dual-energy CT for the diagnosis of gout: an accuracy and diagnostic yield study. Ann Rheum Dis. 2015 Jun;74(6):1072-7. doi: 10.1136/annrheumdis-2013-205095. Epub 2014 Mar 25. PMID 24671771
- [Background] Hidas G, Eliahou R, Duvdevani M, Coulon P, Lemaitre L, Gofrit ON, Pode D, Sosna J. Determination of renal stone composition with dual-energy CT: in vivo analysis and comparison with x-ray diffraction. Radiology. 2010 Nov;257(2):394-401. doi: 10.1148/radiol.10100249. Epub 2010 Aug 31. PMID 20807846
- [Background] Esquivel A, Ferrero A, Mileto A, Baffour F, Horst K, Rajiah PS, Inoue A, Leng S, McCollough C, Fletcher JG. Photon-Counting Detector CT: Key Points Radiologists Should Know. Korean J Radiol. 2022 Sep;23(9):854-865. doi: 10.3348/kjr.2022.0377. PMID 36047540
- [Background] Marcus RP, Fletcher JG, Ferrero A, Leng S, Halaweish AF, Gutjahr R, Vrtiska TJ, Wells ML, Enders FT, McCollough CH. Detection and Characterization of Renal Stones by Using Photon-Counting-based CT. Radiology. 2018 Nov;289(2):436-442. doi: 10.1148/radiol.2018180126. Epub 2018 Aug 7. PMID 30084728
- [Background] Tenforde AS, Fredericson M. Influence of sports participation on bone health in the young athlete: a review of the literature. PM R. 2011 Sep;3(9):861-7. doi: 10.1016/j.pmrj.2011.05.019. PMID 21944303
- [Background] Grunz JP, Heidenreich JF, Lennartz S, Weighardt JP, Bley TA, Ergun S, Petritsch B, Huflage H. Spectral Shaping Via Tin Prefiltration in Ultra-High-Resolution Photon-Counting and Energy-Integrating Detector CT of the Temporal Bone. Invest Radiol. 2022 Dec 1;57(12):819-825. doi: 10.1097/RLI.0000000000000901. Epub 2022 Jun 24. PMID 35776435
- [Background] Grunz JP, Petritsch B, Luetkens KS, Kunz AS, Lennartz S, Ergun S, Bley TA, Huflage H. Ultra-Low-Dose Photon-Counting CT Imaging of the Paranasal Sinus With Tin Prefiltration: How Low Can We Go? Invest Radiol. 2022 Nov 1;57(11):728-733. doi: 10.1097/RLI.0000000000000887. Epub 2022 May 6. PMID 35703452
- See also: Report on the use of patient shielding in radiological procedures Swiss Society of Radiobiology and Medical Physics. — https://ssrpm.ch/wp-content/uploads/2021/01/Report-21.pdf